CLINICAL TRIAL: NCT00379639
Title: A Phase I/II Study of Romidepsin (Depsipeptide) in Combination With Gemcitabine in Patients With Pancreatic and Other Advanced Solid Tumors.
Brief Title: A Study of Romidepsin (Depsipeptide) in Combination With Gemcitabine in Patients With Pancreatic and Other Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GPI-06-0003
Record Dates: First submitted 2006-09-20; First posted 2006-09-22 (Estimated); Results first posted 2012-08-13 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; advanced solid tumors
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — romidepsin; Depsipeptides; Gemcitabine

ARMS (1):
- Romidepsin / Gemcitabine (Experimental): Participants were to receive 7, 10 or 12 mg/m^2 of romidepsin intravenously on either Days 1, 8 and 15 (Schedule A) or Days 1 and 15 (Schedule B) of each 28-day cycle, followed by 800 or 1000 mg/m^2 of gemcitabine. Subsequent doses of both drugs were based on treatment-related toxicities. The planned duration of study therapy was 6 cycles or until disease progression occurred. Patients who responded could continue beyond 6 cycles until disease progression or until a withdrawal criterion was met.
  Interventions: Drug: Romidepsin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Romidepsin — 7, 10 or 12 mg/m^2 via intravenous infusion over 4 hours on either Days 1, 8 and 15 or Days 1 and 15 of each 28-day cycle.
  Other Names: ISTODAX®; Depsipeptide; FK228
Drug: Gemcitabine — 800 or 1000 mg/m^2 via intravenous infusion over 30 minutes on either Days 1,8 and 15 or Days 1 and 15 of each 28 day cycle.
  Other Names: Gemzar®

SUMMARY:
This was a phase I dose escalation trial designed to determine the maximum tolerated dose (MTD) for the combination of romidepsin (depsipeptide) and gemcitabine. The study was originally planned as a Phase I/II; however only Phase I of the study was conducted.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed advanced solid tumors
* measurable or evaluable disease
* written informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1

Exclusion Criteria:

* Prior treatment with romidepsin or gemcitabine
* Prior chemotherapy treatment within 3 weeks prior to the first day of treatment or prior treatment with an investigational agent within 4 weeks prior to the first day of treatment. Patients must have recovered from all therapy-related toxicities (Common Terminology Criteria grade ≤ 1)
* Prior radiotherapy within 4 weeks prior to the first day of treatment. Patients who have not fully recovered or whose acute toxicity related to prior radiotherapy has not returned to baseline are ineligible.
* Prior surgery within 3 weeks prior to the first day of treatment, excluding surgical biopsies and port placements
* Concomitant use of any other anti-cancer therapy
* Concomitant use of any investigational agent
* Use of any investigational agent within 4 weeks of study entry
* Any known cardiac abnormalities, including congenital long QT syndrome, QTcF interval >480 milliseconds, myocardial infarction within 12 months of study entry, coronary artery disease (CAD), congestive heart failure (CHF), evidence of cardiac ischemia at screening, known history of sustained ventricular tachycardia (VT), ventricular fibrillation (VF), Torsade de Pointes, or cardiac arrest, hypertrophic cardiomegaly or restrictive cardiomyopathy chronic hypertension, any cardiac arrhythmia requiring anti-arrhythmic medication
* Serum potassium <3.8 mmol/L or serum magnesium <2.0 mg/dL (electrolyte abnormalities can be corrected with supplementation to meet inclusion criteria)
* Concomitant use of drugs that may cause a prolongation of the QTc
* Concomitant use of CYP3A4 inhibitors
* Clinically significant active infection
* Known infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Inadequate bone marrow or other organ function as evidenced by:

  * Hemoglobin <9 g/dL (Transfusions and/or erythropoietin are permitted.)
  * Absolute neutrophil count (ANC) ≤1.5 x 10^9 cells/L
  * Platelet count <100 x 10^9 cells/L or platelet count <75 x 10^9 cells/L if bone marrow disease involvement is documented
  * Total bilirubin >2.0 x upper limit of normal (ULN)
  * Aspartate transaminase/serum glutamic oxaloacetic transaminase (AST/SGOT) and alanine transaminase/serum glutamic pyruvic transaminase (ALT/SGPT) >2.0 x ULN or >3.0 x ULN in the presence of demonstrable liver metastases
  * Serum creatinine >2.0 x ULN
* Patients who are pregnant or breast-feeding
* Any significant medical or psychiatric condition that might prevent the patient from complying with all study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-07-01 (Actual); Primary Completion 2008-07-01 (Actual); Study Completion 2008-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard A. Burris, M.D., Principal Investigator — SCRI Development Innovations, LLC
Locations (1):
- Sarah Cannon Research Institute, Nashville, Tennessee, United States

REFERENCES:
- [Result] Jones SF, Infante JR, Spigel DR, Peacock NW, Thompson DS, Greco FA, McCulloch W, Burris HA 3rd. Phase 1 results from a study of romidepsin in combination with gemcitabine in patients with advanced solid tumors. Cancer Invest. 2012 Jul;30(6):481-6. doi: 10.3109/07357907.2012.675382. Epub 2012 Apr 26. PMID 22536933

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were assigned to 1 of 2 dose schedules concurrently on an every-other-patient basis using a "3+3" dosing scheme: Patients in Schedule A received study treatment Days 1, 8, and 15 and those in Schedule B on Days 1 and 15 of every 28-day cycle. Patients were observed for 28 days before enrollment at the next dose level, based on toxicities.
Groups:
- Dose Level 1: Participants received romidepsin 10 mg/m^2 plus gemcitabine 800 mg/m^2 on Days 1, 8, and 15 every 28 days.
- Dose Level 2: Participants received romidepsin 7 mg/m^2 plus gemcitabine 800 mg/m^2 on Days 1, 8, and 15 every 28 days.
- Dose Level 5: Participants received romidepsin 10 mg/m^2 plus gemcitabine 800 mg/m^2 on Days 1 and 15 every 28 days.
- Dose Level 6: Participants received romidepsin 10 mg/m^2 plus gemcitabine 1000 mg/m^2 on Days 1 and 15 every 28 days.
- Dose Level 8: Participants received romidepsin 12 mg/m^2 plus gemcitabine 800 mg/m^2 on Days 1 and 15 every 28 days.
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 5 | Dose Level 6 | Dose Level 8
Started | 7 (Represents the number of patients who received any amount of study drug.) | 7 (Represents the number of patients who received any amount of study drug.) | 10 (Represents the number of patients who received any amount of study drug.) | 6 (Represents the number of patients who received any amount of study drug.) | 6 (Represents the number of patients who received any amount of study drug.)
Efficacy Evaluable Population | 6 (Completed ≥2 consecutive treatment cycles, had ≥1 efficacy assessment & no major protocol violations) | 7 (Completed ≥2 consecutive treatment cycles, had ≥1 efficacy assessment & no major protocol violations) | 7 (Completed ≥2 consecutive treatment cycles, had ≥1 efficacy assessment & no major protocol violations) | 4 (Completed ≥2 consecutive treatment cycles, had ≥1 efficacy assessment & no major protocol violations) | 3 (Completed ≥2 consecutive treatment cycles, had ≥1 efficacy assessment & no major protocol violations)
Completed 6 Cycles of Therapy | 4 | 2 | 1 | 0 | 0
Completed | 4 (Represents patients who completed the study through Cycle 6) | 2 (Represents patients who completed the study through Cycle 6) | 1 (Represents patients who completed the study through Cycle 6) | 0 (Represents patients who completed the study through Cycle 6) | 0 (Represents patients who completed the study through Cycle 6)
Not Completed | 3 | 5 | 9 | 6 | 6
Not completed — Disease Progression | 3 | 3 | 3 | 4 | 4
Not completed — Physician Decision | 0 | 2 | 1 | 1 | 0
Not completed — Symptomatic Deterioration | 0 | 0 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 5 | Dose Level 6 | Dose Level 8 | Total
Number analyzed (Participants) | 7 | 7 | 10 | 6 | 6 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (11.25) | 53.4 (11.04) | 62.6 (10.86) | 57.3 (15.54) | 57.0 (13.37) | 58.3 (11.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 4 | 6 | 5 | 25
  Male | 2 | 2 | 6 | 0 | 1 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 7 | 10 | 6 | 6 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 6 | 6 | 10 | 6 | 6 | 34
  Black | 1 | 0 | 0 | 0 | 0 | 1
  Pakistani | 0 | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 10 | 6 | 6 | 36
Height [Mean (Standard Deviation); unit: cm] | 169.3 (9.52) | 163.7 (8.13) | 170.9 (10.33) | 159.6 (4.09) | 164.9 (8.71) | 166.3 (9.21)
Weight [Mean (Standard Deviation); unit: kg] | 79.8 (20.54) | 77.6 (25.21) | 73.1 (12.58) | 69.0 (26.84) | 61.7 (27.56) | 72.7 (21.70)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] | 1.9 (0.28) | 1.8 (0.29) | 1.8 (0.19) | 1.7 (0.23) | 1.7 (0.35) | 1.8 (0.27)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Dose-limiting Toxicity (DLT)
Description: Toxicities were assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), V 3.0. A DLT was one of the following, if considered at least possibly related to study treatment:
  Grade 4 neutropenia for ≥5 days or febrile neutropenia; Grade 4 thrombocytopenia or need for a platelet transfusion; ≥ Grade 3 nausea and/or emesis despite using optimal antiemetic therapy; ≥ Grade 3 diarrhea despite using maximal supportive therapy; Any clinically significant Grade 3 or 4 nonhematologic toxicity; Inability to administer all doses in cycle 1.
Time Frame: 28 days
Population: Safety population - all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 5 | Dose Level 6 | Dose Level 8
Number analyzed (Participants) | 7 | 7 | 10 | 6 | 6
participants | 3 | 1 | 0 | 2 | 0

2. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: AEs were graded for severity according to the National Cancer Institute Common Terminology Criteria (NCI CTCAE), V 3.0: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe (prevents normal everyday activities); Grade 4: Life-threatening or disabling; Grade 5: Death.
  A serious AE is associated with events that pose a threat to a patient's life or functioning, require hospitalization, is a congenital anomaly/birth defect or is an important medical event or condition that may jeopardize the patient and may require medical or surgical intervention to prevent one of the above outcomes.
Time Frame: From the date of first dose to 30 days after last dose (up to 236 days).
Population: Safety population.
Measure: Number; unit: participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 5 | Dose Level 6 | Dose Level 8
Number analyzed (Participants) | 7 | 7 | 10 | 6 | 6
participants
  Any adverse event | 7 | 7 | 10 | 6 | 6
  ≥Grade 3 adverse event | 7 | 5 | 5 | 4 | 3
  Grade 4 adverse event | 1 | 2 | 3 | 2 | 1
  Serious adverse event | 3 | 2 | 4 | 1 | 2
  Adverse event leading to discontinuation | 0 | 0 | 1 | 0 | 1
  Adverse event leading to death | 0 | 0 | 0 | 0 | 1

3. Primary Outcome: Best Overall Response
Description: Disease response was determined by the Investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria using computed tomography or magnetic resonance imaging:
  Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions; Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions or the appearance of ≥1 new lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Disease assessments were performed within 4 weeks of first dose and every 8 weeks thereafter (up to 236 days).
Population: The Efficacy Evaluable (EE) population consisted of all patients who completed at least 2 consecutive cycles of treatment, had at least 1 post-Baseline efficacy assessment performed, and did not have any major protocol violations.
Measure: Number; unit: participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 5 | Dose Level 6 | Dose Level 8
Number analyzed (Participants) | 6 | 7 | 7 | 4 | 3
participants
  Complete Response | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 1 | 0 | 0 | 1
  Stable disease | 5 | 4 | 3 | 1 | 1
  Progressive disease | 1 | 2 | 4 | 3 | 1

ADVERSE EVENTS:
Time Frame: From the date of first dose to 30 days after last dose.
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 5 | Dose Level 6 | Dose Level 8
Serious Adverse Events (participants affected / at risk) | 3/7 | 2/7 | 4/10 | 1/6 | 2/6
Other Adverse Events (participants affected / at risk) | 7/7 | 7/7 | 10/10 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=7) | Dose Level 2 (N=7) | Dose Level 5 (N=10) | Dose Level 6 (N=6) | Dose Level 8 (N=6)
Anaemia NOS (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain NOS (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0
Small intestinal obstruction NOS (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting NOS (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Pneumonia NOS (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=7) | Dose Level 2 (N=7) | Dose Level 5 (N=10) | Dose Level 6 (N=6) | Dose Level 8 (N=6)
Anaemia NOS (Blood and lymphatic system disorders) | 3 | 2 | 1 | 2 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 4 | 1 | 4 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Abdominal pain NOS (Gastrointestinal disorders) | 4 | 3 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 5 | 5 | 3 | 3
Diarrhoea NOS (Gastrointestinal disorders) | 1 | 3 | 2 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 7 | 7 | 5 | 4
Reflux oesophagitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Vomiting NOS (Gastrointestinal disorders) | 5 | 5 | 7 | 5 | 5
Asthenia (General disorders) | 2 | 0 | 2 | 1 | 1
Chest pain (General disorders) | 0 | 3 | 2 | 0 | 0
Fatigue (General disorders) | 6 | 6 | 9 | 4 | 1
Oedema peripheral (General disorders) | 0 | 1 | 1 | 0 | 0
Pain NOS (General disorders) | 3 | 2 | 1 | 0 | 0
Performance status decreased (General disorders) | 0 | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 3 | 0 | 1 | 1
Urinary tract infection NOS (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 2 | 1 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 4 | 7 | 4 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2 | 3 | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 0 | 3
Dysgeusia (Nervous system disorders) | 1 | 1 | 4 | 2 | 1
Headache (Nervous system disorders) | 2 | 0 | 2 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 1 | 2 | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Rash NOS (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 1 | 0
Hypertension NOS (Vascular disorders) | 0 | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Upon investigator submission of a publication or presentation to Celgene, Celgene shall complete its review within 60 days after receipt of the proposed publication or presentation. Upon Celgene's request, proposed publication or presentation will be delayed up to 60 additional days to enable Celgene to secure adequate intellectual property protection of property of Celgene that would be affected by such proposed publication or presentation